CLINICAL TRIAL: NCT02871089
Title: An Open-label, Multicentre, Randomised, Single-period, Parallel Design Study to Assess the Effect of Closed Loop Insulin Delivery From Onset of Type 1 Diabetes in Youth on Residual Beta Cell Function Compared to Standard Insulin Therapy
Brief Title: Closed Loop From Onset in Type 1 Diabetes
Acronym: CLOuD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); Alder Hey Children's NHS Foundation Trust (Other); Nottingham University Hospitals NHS Trust (Other); Oxford University Hospitals NHS Trust (Other); University Hospital Southampton NHS Foundation Trust (Other); Jaeb Center for Health Research (Other); The Leeds Teaching Hospitals NHS Trust (Other); University of Edinburgh (Other)
Responsible Party: Principal Investigator, Dr Roman Hovorka, Director of Research, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CLOuD
Record Dates: First submitted 2016-07-27; First posted 2016-08-18 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus; Type 1 Diabetes
Keywords: Type 1 Diabetes; Closed-loop glucose control; Artificial Pancreas; Continuous subcutaneous insulin infusion; Multiple daily injection therapy; New onset type 1 diabetes; Residual C-Peptide secretion; Beta-cell function preservation; Continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 24/7 Closed loop delivery (Experimental): Unsupervised home use of day and night automated closed-loop insulin delivery system FlorenceM (Medtronic 640G insulin pump, guardian 3 CGM and Android smartphone) of CamAPS FX (Dana insulin pump, Dexcom G6 CGM and App on Android smartphone) until 24 months after diagnosis
  Interventions: Device: Closed-loop system (Florence M or CamAPS FX)
- Multiple Daily Injections (Active Comparator): Participants will apply standard insulin therapy using multiple daily injections via insulin pens during the 24 months control period
  Interventions: Other: Multiple Daily Injections

INTERVENTIONS:
Device: Closed-loop system (Florence M or CamAPS FX) — The automated closed-loop system (FlorenceM) will consist of:
  * Sensor augmented Medtronic insulin pump 640G (Medtronic Minimed, CA, USA) incorporating the Medtronic Enlite/Guardian 3 real time CGM and glucose suspend feature.
  * An Android smartphone containing the Cambridge model predictive algorithm and communicating wirelessly with the insulin pump using a proprietary translator device.
  The automated closed-loop system (CamAPS FX) will consist of:
  * Dana R or RS insulin pump
  * Dexcom G6 real-time CGM
  * CamAPS FX App on an unlocked android smartphone.
  Rapid acting insulin analogue will be used (insulin aspart, insulin lispro, insulin glulisine or similar or ultra-rapid insulin analogue).
  Arms: 24/7 Closed loop delivery
Other: Multiple Daily Injections — Rapid acting insulin analogue and long acting insulin analogue will be subcutaneously administered using CE-marked insulin pen devices in accordance with the manufacturer's instructions for their intended purposes.
  Participants will be given long acting analogue (insulin glargine, insulin detemir or similar) once or twice daily according to their needs and boluses of rapid acting analogue (insulin aspart, insulin lispro, insulin glulisine or similar or ultra-rapid insulin analogue) when carbohydrates are consumed.
  Arms: Multiple Daily Injections

SUMMARY:
The purpose of the study is to use a novel treatment approach, the artificial pancreas, after diagnosis of type 1 diabetes (T1D) to improve glucose control with the anticipated improvements of residual C-peptide secretion.

This is an open-label, multicentre, single-period, randomised, parallel group design study. It is expected that a total of up to 190 subjects (aiming for 96 randomised subjects) will be recruited within ten working days of diagnosis of type 1 diabetes through paediatric diabetes centres in the UK. Half of the participants aged 10 to 16.9 years will be treated by conventional insulin injections and the other half by the artificial pancreas (closed loop insulin delivery system). Each treatment will last 24 months. All participants completing the 24 month study period will be invited to continue in an optional extension phase with the treatment allocated at randomisation for a further 24 months.

Subjects in the intervention group will receive additional training on components of the artificial pancreas, i.e. insulin pump and continuous glucose monitoring (CGM), prior to starting closed loop insulin delivery. Subjects in the control intervention group will continue with standard therapy, i.e. multiple daily injection therapy. The study includes up to 14 visits and 1 telephone/email contact for subjects completing the study. After run-in and randomisation, visits will be conducted every 3 months in both arms. Beta-cell function will be assessed by serial measurement of C-peptide in response to a standardised mixed meal tolerance test (MMTT). MMTTs will be conducted at baseline, 6-,12- and 24 months post diagnosis.

The primary outcome is the between group difference in the area under the stimulated C-peptide curve (AUC) of the MMTT at 12 month post diagnosis. Secondary outcomes include between group differences in stimulated C-peptide AUC over 24 months, differences in glycaemic control as assessed by HbA1c, time spent in glucose target range, glucose variability, hypo- and hyperglycaemia as recorded by periodically applied CGM, as well as insulin requirements and change in bodyweight. Additionally, cognitive, emotional and behavioural characteristics of participating subjects and parents will be assessed, and a cost utility analysis on the benefits of closed loop insulin delivery will be performed. Safety evaluation comprises assessment of the frequency of severe hypoglycaemic episodes, diabetic ketoacidosis (DKA) and number, nature and severity of other adverse events.

DETAILED DESCRIPTION:
Purpose of the study:

* To determine whether continued intensive metabolic control using closed loop insulin delivery (CL) following diagnosis of type 1 diabetes can preserve C-peptide secretion as a marker of residual beta cell function compared to standard multiple daily injections (MDI) therapy

Primary objective:

* To assess residual C-peptide secretion 12 months after diagnosis of type 1 diabetes in participants receiving either CL insulin delivery or standard MDI therapy

Secondary Objectives:

* Biochemical:

  * To compare effects of study interventions on residual C-peptide secretion over 24 months following diagnosis
  * To examine how intensive diabetes management using CL insulin delivery affects glucose control in terms of safety and efficacy over 24 months
* Human Factors: To assess cognitive, emotional, and behavioural characteristics of participating subjects and family members and their response to closed loop insulin delivery and clinical trial
* Health economics: To perform cost utility analysis and inform reimbursement decision-making

Study design:

* An open-label, multi-centre, randomised, single period, two-arm parallel group study with internal pilot, contrasting closed loop with MDI with an optional 24 month extension phase.

Sample Size:

* 96 participants randomised (48 per group); each clinical site will aim to recruit between 15 and 20 participants

Maximum duration of study for a subject:

* 24 months (48 months if opting to participate in extension phase)

Recruitment:

* Recruitment will take place at Addenbrooke's Hospital, Cambridge, Leeds Teaching Hospital, Leeds, Alder Hey Children's Hospital, Liverpool, Nottingham Hospital, Nottingham, Oxford Children's Hospital, Oxford, Southampton Children's Hospital, Southampton and Royal Hospital for Sick Children, Edinburgh..

Consent

* Written consent/assent will be obtained from participants and/or guardians according to Research Ethics Committee (REC) requirements.

Screening and baseline assessment:

Eligible participants will undergo a screening evaluation including the following activities:

* medical (diabetes) history
* body weight, height and blood pressure measurement
* record of current insulin therapy
* screening and baseline blood sampling

During a baseline visit, the following assessments/ interventions will be carried out at the clinical research facility:

* mixed meal tolerance test (MMTT)
* blood sampling for lipid profile
* centrally measured HbA1c and subsequent immunological analyses
* questionnaires
* computerised cognitive testing
* initiating blinded CGM to assess baseline glycaemic control

Run in period:

* Following consent/screening and baseline assessment, multiple daily injection therapy will be continued in all participants. All participants will receive non study related core diabetes training as per usual clinical practice for a period of up to three weeks.
* All subjects will be provided with 24 hour telephone helpline and will also be given written instructions about when to contact clinical team.

Randomisation:

* Eligible participants will be randomised in a 1:1 ratio using central randomisation software to either closed loop or standard therapy i.e. MDI.

  1. Closed loop (interventional arm) Following randomisation, participants in the closed loop group will receive additional training sessions to cover key aspects of insulin pump use and CGM, prior to starting closed loop insulin delivery.

     Once competent in the use of the study pump and CGM system, participants will receive training required for safe and effective use of the closed loop system. During a 2-4 hour session participants will operate the system under the supervision of the clinical team. Competency on the use of closed loop system will be evaluated. Thereafter, participants are expected to use closed loop for 24 months without supervision or remote monitoring. The 24 hour support helpline will be available in case of problems.
  2. Multiple daily injections (control arm) Participants in the control group will receive additional training sessions following randomisation including a refresher on carbohydrate counting skills, and insulin dose adjustments.

Standard therapy (i.e. MDI) will be applied for 24 months. Participants will be allowed to switch to insulin pump therapy if clinically indicated.

Follow up assessments (3-, 6-, 9-, 12-, 15-, 18-, 21- months):

* Follow up study visits will be conducted 3 monthly including data downloads/recording of insulin requirements, adverse event recording, and blood sampling (HbA1c).
* Participants will be fitted with blinded CGM systems at the end of each follow up visit. The sensors will be worn at home for up to 14 days and will be sent back to the research team.
* MMTTs will be performed at 6 month and 12 month follow up visit.
* Sleep will be assessed using a wristwatch device for 7 days following study visits at 6 and 12 months post diagnosis. Concomitantly, a sleep diary and sleep quality questionnaire will be distributed.
* Validated questionnaires evaluating the impact of the technology on quality of life, life change, diabetes management and fear of hypoglycaemia will be completed at the 12 month visit.
* At 12 months, participants will repeat the computerised cognitive tests first administered at baseline.
* Qualitative interviews will be conducted at month 12 in a subset of subjects and parents int he closed-loop arm.

End of study assessments (24 months):

* A MMTT will be performed.
* A blood sample will be taken for measurement of HbA1c, lipids and immunological analyses.
* Validated questionnaires evaluating the impact of the technology on quality of life, life change, diabetes management and fear of hypoglycaemia will be completed.
* Participants will repeat the computerised cognitive tests first administered at baseline.
* Sleep will be assessed using a wristwatch device for 7 days within the last month of the trial. Concomitantly, a sleep diary and sleep quality questionnaire will be distributed.
* Participants and families will be invited to attend focus group discussions. 24-hour telephone helpline:
* In case of any technical device or problems related to diabetes management such as hypo- or hyperglycaemia, subjects will be able to contact a 24-hour telephone helpline to the local clinical and research team at any time. The local research team will have access to central 24 hour advice on technical issues.

Procedures for safety monitoring during trial:

* Standard operating procedures for monitoring and reporting of all adverse events (AE) will be in place, including serious adverse events (SAE), serious adverse device effects (SADE) and specific adverse events such as severe hypoglycaemia.
* Subjects will be asked to test and record blood or urine ketones if their finger prick glucose is above 14.0 mmol/l, as part of the safety assessment for hyperglycaemia.
* A data monitoring and ethics committee (DMEC) will be informed of all serious adverse events and any unanticipated serious adverse device effects that occur during the study and will review compiled adverse event data at periodic intervals.

Criteria for withdrawal of patients on safety grounds:

* A subject, parent, or guardian may terminate participation in the study at any time without necessarily giving a reason and without any personal disadvantage. An investigator can stop the participation of a subject after consideration of the benefit/risk ratio. Possible reasons are:

  1. Serious adverse events
  2. Significant protocol violation or non-compliance
  3. Failure to satisfy competency assessment
  4. Decision by the investigator, or the Sponsor, that termination is in the subject's best medical interest
  5. Pregnancy, planned pregnancy, or breast feeding
  6. Allergic reaction to insulin Efforts will be made to retain subjects in follow up for the final primary outcome assessment even if the intervention is discontinued, unless the investigator believes that it will be harmful for the subject to continue in the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of type 1 diabetes within previous 21 days. Day 1 will be defined as the day insulin was first administered. Type 1 diabetes will be defined according to WHO criteria using standard diagnostic practice.

   [WHO definition: 'The aetiological type named type 1 encompasses the majority of cases with are primarily due to beta-cell destruction, and are prone to ketoacidosis. Type 1 includes those cases attributable to an autoimmune process, as well as those with beta-cell destruction for which neither an aetiology nor a pathogenesis is known (idiopathic). It does not include those forms of beta-cell destruction or failure to which specific causes can be assigned (e.g. cystic fibrosis, mitochondrial defects, etc.).']
2. The subject is at least 10 years and not older than 16.9 years
3. The subject/carer is willing to perform regular capillary blood glucose monitoring, with at least 4 blood glucose measurements taken every day
4. The subject is literate in English
5. The subject is willing to wear glucose sensor
6. The subject is willing to wear closed loop system at home
7. The subject is willing to follow study specific instructions
8. The subject is willing to upload pump and CGM data at regular intervals

Exclusion Criteria:

1. Physical or psychological condition likely to interfere with the normal conduct of the study and interpretation of the study results as judged by the investigator
2. Current treatment with drugs known to interfere with glucose metabolism, e.g. systemic corticosteroids, non-selective beta-blockers and MAO inhibitors etc.
3. Known or suspected allergy to insulin
4. Regular use of acetaminophen
5. Lack of reliable telephone facility for contact
6. Pregnancy, planned pregnancy, or breast feeding
7. Living alone
8. Severe visual impairment
9. Severe hearing impairment
10. Medically documented allergy towards the adhesive (glue) of plasters or unable to tolerate tape adhesive in the area of sensor placement
11. Serious skin diseases (e.g. psoriasis vulgaris, bacterial skin diseases) located at places of the body, which potentially are possible to be used for localisation of the glucose sensor
12. Illicit drugs abuse
13. Prescription drugs abuse
14. Alcohol abuse
15. Sickle cell disease, haemoglobinopathy, receiving red blood cell transfusion or erythropoietin within 3 months prior to time of screening
16. Eating disorder such as anorexia or bulimia
17. Milk protein allergy

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Area under the meal stimulated C-peptide curve (AUC) during a mixed meal tolerance test (MMTT) | 12 months post diagnosis

SECONDARY OUTCOMES:
Mean stimulated C-peptide AUC during a mixed meal tolerance test | Baseline, 6 months and 24 months post diagnosis
HbA1c Levels | Baseline, 3, 6, 9, 12, 15, 18, 21 and 24 months post diagnosis
  Both arms
Percentage of patients in each group with HbA1c <7.5% (58mmol/mol) | Baseline, 3, 6, 9, 12, 15, 18, 21 and 24 months post diagnosis
  Both arms
Percentage of time spent with sensor glucose readings in the target range (3.9 to 10mmol/l) | Baseline, 3, 6, 9, 12, 15, 18, 21 and 24 months post diagnosis
  Both arms
Mean sensor glucose level | Baseline, 3, 6, 9, 12, 15, 18, 21 and 24 months post diagnosis
  Both arms
Standard deviation of sensor glucose levels | Baseline, 3, 6, 9, 12, 15, 18, 21 and 24 months post diagnosis
  Both arms
Coefficient of variation of sensor levels | Baseline, 3, 6, 9, 12, 15, 18, 21 and 24 months post diagnosis
  Both arms
Percentage of time with sensor glucose levels <3.5 mmol/l and <2.8 mmol/l | Baseline, 3, 6, 9, 12, 15, 18, 21 and 24 months post diagnosis
  Both arms
Percentage of time spent below target glucose (3.9mmol/l) | Baseline, 3, 6, 9, 12, 15, 18, 21 and 24 months post diagnosis
  Both arms
AUC of sensor glucose below 3.5mmol/l | Baseline, 3, 6, 9, 12, 15, 18, 21 and 24 months post diagnosis
  Both arms
Time spent with sensor glucose above target (10.0 mmol/l) | Baseline, 3, 6, 9, 12, 15, 18, 21 and 24 months post diagnosis
  Both arms
Time with sensor glucose levels in significant hyperglycaemia (glucose levels > 16.7 mmol/l) | Baseline, 3, 6, 9, 12, 15, 18, 21 and 24 months post diagnosis
  Both arms
Insulin Requirements | Baseline, 3, 6, 9, 12, 15, 18, 21 and 24 months post diagnosis
  Total, basal and bolus insulin dose (U/kg). Both arms
Weight | Baseline, 6, 12 and 24 months post diagnosis
  Change in body mass index (BMI) standard deviation score. Both arms
Blood pressure | Baseline, 6, 12 and 24 months post diagnosis
  Both arms
Lipid profile | Baseline, 12 and 24 months post diagnosis
  Both arms

OTHER OUTCOMES:
Severe hypoglycaemic episodes | 24 month intervention period
  Frequency of severe hypoglycaemic episodes
Diabetes ketoacidosis | 24 month intervention period
  Frequency of severe diabetes ketoacidosis
Adverse Events | 24 month intervention period + 3 weeks
  Number, nature and severity of other adverse events. The period during which adverse events will be reported is defined as the period from the beginning of the study (obtaining informed consent) until 3 weeks after the end of the study participation
Serious Adverse Events | 24 month intervention period + 3 weeks
  Number, nature and severity of serious adverse events. The period during which adverse events will be reported is defined as the period from the beginning of the study (obtaining informed consent) until 3 weeks after the end of the study participation
Assessment of the frequency of use of the closed loop system | 24 month intervention period
  Utility evaluation
Assessment of the duration of use of the closed loop system. | 24 month intervention period
  Utility evaluation
Cognitive Assessment | Baseline, 6, 12 and 24 months post diagnosis
  Assessment of cognitive changes using computerized cognitive testing.
Health Economic Evaluation | 24 month intervention period
  Cost utility analysis using the CORE Diabetes Model (CDM; IMS Health, Basel, Switzerland) on the benefits of closed loop insulin delivery to inform reimbursement decision-making.
Quantitative Human Factor Assessment | Baseline,12 and 24 months post diagnosis
  Questionnaires will be completed by participants and parents/guardians.
Qualitative Human Factor Assessment | 12 and 24 months post diagnosis
  Interview and focus group with participants and parents/guardians.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Hovorka, PhD, Study Director — Department of Paediatrics, University of Cambridge, UK; Ajay Thankamony, MD, Principal Investigator — Department of Paediatrics, University of Cambridge, UK; Atrayee Ghatak, MD, Principal Investigator — Alder Hey Children's NHS Foundation Trust, Liverpool; Tabitha Randell, MD, Principal Investigator — Nottingham Children's Hospital, Nottingham, UK; Rachel Besser, MD, Principal Investigator — Oxford Children's Hospital, Oxford, UK; Nicola Trevelyan, MD, Principal Investigator — Southampton Children's Hospital, Southampton, UK; Daniela Elleri, MD, Principal Investigator — Royal Hospital for Sick Children, Edinburgh, UK; Fiona Campbell, MD, Principal Investigator — Leeds Children's Hospital
Locations (7):
- United Kingdom (7):
  - Southampton Children's Hospital, Southampton, Hampshire
  - Nottingham Children's Hospital, Nottingham, Nottinghamshire
  - John Radcliffe Hospital, Oxford, Oxfordshire
  - Alder Hey Children's NHS Foundation Trust, Liverpool, West Derby
  - St James's University Hospital, Leeds, West Yorkshire
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Royal Hospital for Sick Children, Edinburgh

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Hovorka R. Artificial Pancreas Project at Cambridge 2013. Diabet Med. 2015 Aug;32(8):987-92. doi: 10.1111/dme.12766. Epub 2015 Apr 15. PMID 25819473
- [Background] Thabit H, Tauschmann M, Allen JM, Leelarathna L, Hartnell S, Wilinska ME, Acerini CL, Dellweg S, Benesch C, Heinemann L, Mader JK, Holzer M, Kojzar H, Exall J, Yong J, Pichierri J, Barnard KD, Kollman C, Cheng P, Hindmarsh PC, Campbell FM, Arnolds S, Pieber TR, Evans ML, Dunger DB, Hovorka R. Home Use of an Artificial Beta Cell in Type 1 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2129-2140. doi: 10.1056/NEJMoa1509351. Epub 2015 Sep 17. PMID 26379095
- [Background] Tauschmann M, Allen JM, Wilinska ME, Thabit H, Stewart Z, Cheng P, Kollman C, Acerini CL, Dunger DB, Hovorka R. Day-and-Night Hybrid Closed-Loop Insulin Delivery in Adolescents With Type 1 Diabetes: A Free-Living, Randomized Clinical Trial. Diabetes Care. 2016 Jul;39(7):1168-74. doi: 10.2337/dc15-2078. Epub 2016 Jan 6. PMID 26740634
- [Derived] Boughton CK, Allen JM, Ware J, Wilinska ME, Hartnell S, Thankamony A, Randell T, Ghatak A, Besser REJ, Elleri D, Trevelyan N, Campbell FM, Sibayan J, Calhoun P, Bailey R, Dunseath G, Hovorka R; CLOuD Consortium. Closed-Loop Therapy and Preservation of C-Peptide Secretion in Type 1 Diabetes. N Engl J Med. 2022 Sep 8;387(10):882-893. doi: 10.1056/NEJMoa2203496. PMID 36069870
- [Derived] Rankin D, Kimbell B, Allen JM, Besser REJ, Boughton CK, Campbell F, Elleri D, Fuchs J, Ghatak A, Randell T, Thankamony A, Trevelyan N, Wilinska ME, Hovorka R, Lawton J. Adolescents' Experiences of Using a Smartphone Application Hosting a Closed-loop Algorithm to Manage Type 1 Diabetes in Everyday Life: Qualitative Study. J Diabetes Sci Technol. 2021 Sep;15(5):1042-1051. doi: 10.1177/1932296821994201. Epub 2021 Jul 14. PMID 34261348
- [Derived] Rankin D, Kimbell B, Hovorka R, Lawton J. Adolescents' and their parents' experiences of using a closed-loop system to manage type 1 diabetes in everyday life: qualitative study. Chronic Illn. 2022 Dec;18(4):742-756. doi: 10.1177/1742395320985924. Epub 2021 Jan 20. PMID 33472409
- [Derived] Boughton C, Allen JM, Tauschmann M, Hartnell S, Wilinska ME, Musolino G, Acerini CL, Dunger PD, Campbell F, Ghatak A, Randell T, Besser R, Trevelyan N, Elleri D, Northam E, Hood K, Scott E, Lawton J, Roze S, Sibayan J, Kollman C, Cohen N, Todd J, Hovorka R; CLOuD Consortium. Assessing the effect of closed-loop insulin delivery from onset of type 1 diabetes in youth on residual beta-cell function compared to standard insulin therapy (CLOuD study): a randomised parallel study protocol. BMJ Open. 2020 Mar 12;10(3):e033500. doi: 10.1136/bmjopen-2019-033500. PMID 32169925